CLINICAL TRIAL: NCT04137471
Title: Ontological Addiction Scale: Study Protocol for Scale Validation
Brief Title: Validation of the Ontological Addiction Scale
Acronym: OAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0466
Record Dates: First submitted 2019-09-30; First posted 2019-10-24 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Mood Disorders; Emotional Disorder
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

Bypassing a reductionist view of existing diagnostic categories, ontological addiction theory (OAT) is a new psychological model of human functioning and mental illness. Ontological addiction is a maladaptive condition that stems from an erroneous belief in an inherently existing Self or "I", which is deemed to be the root of all suffering. Five experts from four different countries have created the Ontological Addiction Scale (OAS) to measure the condition and its impact on people's lives. The purpose of this study is to test this scale, evaluating levels of ontological addiction in individuals suffering from emotional or mood disorder, and assess its psychometric properties.

Methods:

This trial will be conducted in compliance with the COSMIN Guidelines. The investigators will collect data from 400 individuals, aged 18 to 70, suffering from emotional or mood disorder, referred to the Therapeutic Center for Mood and Emotional Disorders for an 8-week-mindfulness-based-intervention. Patients will complete the OAS at three time points: one month before the beginning of the therapy, within one week prior to the beginning of therapy, and one year after the end of the therapy. This scale will be completed in conjunction with other practice assessments relating to the psychotherapeutic program. The psychometric properties of the OAS will be assessed.

Discussion:

The Investigators aim to validate a scale assessing a psychological dimension as the root of all mental disorders. The present study may contribute to overcoming limitations of categorical understanding of mental disorders, thus moving toward a more encompassing dimensional comprehension. The scale is responsive to current thinking in modern psychiatry, and it is envisaged that its validation will deeply impact research and care perspectives

ELIGIBILITY:
Inclusion criteria:

An individual must fulfill all of the following criteria in order to be eligible for study enrollment:

* Aged between 18 and 70 years
* Suffering from mood disorder (bipolar or unipolar) and/or emotional disorder (subjective complaint for difficulties to regulate emotions).
* Being referred to the Therapeutic Center for Mood and Emotional Disorders for an 8-week-mindfulness-based-intervention
* Subjects must be able to attend all scheduled visits and to comply with all trial procedures
* Subjects must be covered by public health insurance

Exclusion criteria

* Subject unable to read or/and write
* Psychosis
* Subject who are in a dependency or employment with the sponsor or the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individual suffering from mood disorder (bipolar or unipolar) and/or emotional disorder (subjective complaint for difficulties to regulate emotions).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Validation of the Ontological Addiction Scale by measurement of its psychometric properties | one year after the end of the therapy
  Evaluation of the structural validity of the Ontological Addiction Scale (OAS)

SECONDARY OUTCOMES:
Measurement of the structural validity of the Ontological Addiction Scale by means of factor analysis (the technique of rotation of the main axes varimax will be used) | pre-treatment (first assessment) within one week prior to the beginning of therapy
  Evaluation of the structural validity of the Ontological Addiction Scale (OAS)
Measurement of internal consistency of the Ontological Addiction Scale by a multitrait analysis (assessment of redundancy between items, validation of item consistency, assessment of item dimension intercorrelations) | pre-treatment (first assessment) within one week prior to the beginning of therapy
  Evaluation of internal consistency of the Ontological Addiction Scale (OAS)
Measurement of reliability of the Ontological Addiction Scale by test-retest (degree to which the measurement is free from measurement error) | pre-treatment (first assessment) within one week prior to the beginning of therapy
  Evaluation of reliability of the Ontological Addiction Scale (OAS)
Error measurement of the Ontological Addiction Scale by the calculation of the Strandard Error of the Mean. | pre-treatment (first assessment) within one week prior to the beginning of therapy
  Measurment error of the Ontological Addiction Scale (OAS)
Content validity measurement of the Ontological Addiction Scale | pre-treatment (first assessment) within one week prior to the beginning of therapy
  Content validity measurement of the Addiction Scale (OAS) by content validity index (assessment of the simplicity and clarity of the questionnaire on a 4-point likert scale from not relevant to highly relevant. The answers will then be dichotomized as "not relevant" (score 1 or 2) or "relevant" (score 3 or 4)).
Levels of concern about the mental representation that patients have of themselves (ontological addiction) by the Ontological Addiction Scale (by responding either "never", "rarely", "sometimes", "often", "always" to the 24 items) | pre-treatment (first assessment) within one week prior to the beginning of therapy
  Evaluation of ontological addiction by the ontological addiction scale
Measurement of the structural validity of the Ontological Addiction Scale by means of factor analysis (the technique of rotation of the main axes varimax will be used) | post therapy (second assessment) within the week following completion of therapy
  Evaluation of the structural validity of the Ontological Addiction Scale (OAS)
Measurement of internal consistency of the Ontological Addiction Scale by a multitrait analysis (assessment of redundancy between items, validation of item consistency, assessment of item dimension intercorrelations) | post therapy (second assessment) within the week following completion of therapy
  Evaluation of internal consistency of the Ontological Addiction Scale (OAS)
Measurement of reliability of the Ontological Addiction Scale by test-retest (degree to which the measurement is free from measurement error) | post therapy (second assessment) within the week following completion of therapy
  Evaluation of reliability of the Ontological Addiction Scale (OAS)
Error measurement of the Ontological Addiction Scale by the calculation of the Strandard Error of the Mean | post therapy (second assessment) within the week following completion of therapy
  Measurment error of the Ontological Addiction Scale (OAS)
Content validity measurement of the Ontological Addiction Scale | post therapy (second assessment) within the week following completion of therapy
  Content validity measurement of the Addiction Scale (OAS) by content validity index (assessment of the simplicity and clarity of the questionnaire on a 4-point likert scale from not relevant to highly relevant). The answers will then be dichotomized as "not relevant" (score 1 or 2) or "relevant" (score 3 or 4)).
Levels of concern about the mental representation that patients have of themselves (ontological addiction) by the Ontological Addiction Scale (by responding either "never", "rarely", "sometimes", "often", "always" to the 24 items) | post therapy (second assessment) within the week following completion of therapy
  Evaluation of ontological addiction by the ontological addiction scale
Measurement of the structural validity of the Ontological Addiction Scale by means of factor analysis (the technique of rotation of the main axes varimax will be used) | one year after the end of the therapy.
  Evaluation of the structural validity of the Ontological Addiction Scale (OAS)
Measurement of internal consistency of the Ontological Addiction Scale by a multitrait analysis (assessment of redundancy between items, validation of item consistency, assessment of item dimension intercorrelations) | Evaluation of internal consistency of the Ontological Addiction Scale (OAS)
  one year after the end of the therapy.
Measurement of reliability of the Ontological Addiction Scale by test-retest (degree to which the measurement is free from measurement error) | one year after the end of the therapy.
  Evaluation of reliability of the Ontological Addiction Scale (OAS)
Error measurement of the Ontological Addiction Scale by the calculation of the Strandard Error of the Mean | one year after the end of the therapy.
  Measurment error of the Ontological Addiction Scale (OAS)
Content validity measurement of the Ontological Addiction Scale | one year after the end of the therapy.
  Content validity measurement of the Addiction Scale (OAS) by content validity index (assessment of the simplicity and clarity of the questionnaire on a 4-point likert scale from not relevant to highly relevant). The answers will then be dichotomized as "not relevant" (score 1 or 2) or "relevant" (score 3 or 4)).
Levels of concern about the mental representation that patients have of themselves (ontological addiction) by the Ontological Addiction Scale (by responding either "never", "rarely", "sometimes", "often", "always" to the 24 items) | one year after the end of the therapy.
  Evaluation of ontological addiction by the ontological addiction scale

CONTACTS AND LOCATIONS:
Overall Officials: DEBORAH DUCASSE, MD, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC